CLINICAL TRIAL: NCT06854718
Title: Caregiver-assisted Pain Coping Skills Training for Dementia Pilot Study
Brief Title: Pain With Dementia
Acronym: PWD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute on Aging (NIA) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00116129; 1R61AG088938-01 (NIH)
Record Dates: First submitted 2025-02-10; First posted 2025-03-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-06

CONDITIONS: Pain; Dementia, Mild; Dementia, Moderate
MeSH Terms: conditions — Pain; Dementia; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient-Caregiver Dyads (Other): Patient and caregiver dyads will receive five 45-60 minute sessions over 6-8 week period. This will be over videoconference with a masters-level therapist. All sessions will be audio recorded.
  Interventions: Behavioral: Caregiver-Assisted Pain Coping Skills Training (CG-PCST)

INTERVENTIONS:
Behavioral: Caregiver-Assisted Pain Coping Skills Training (CG-PCST) — Patient-caregiver dyads will receive five, forty-to-sixty-minute sessions over a six-to-eight-week period with a therapist to learn pain coping skills. These include training caregivers in strategies for assessing patient pain, including nonverbal pain behaviors (e.g., grimacing, bodily tension, labored breathing), which will become increasingly important as the patient's ability to express pain verbally decreases. The therapist will also train the caregiver to coach the patient in the use of the skills during activities that are challenging because of pain. We will focus on increasing positive patient-caregiver interactions and patient engagement in valued activities. Throughout the training, the therapist will help the patient and caregiver learn strategies for fostering regular home practice and application of the skills, identify challenges in using the skills, and find strategies for coping with challenges.

SUMMARY:
The purpose of the study is to develop a caregiver-assisted pain coping skills training program for older adults who have pain and mild to moderate dementia and are living at home with a family caregiver. The investigators are planning to recruit 30 patient-caregiver dyads (60 individuals).

DETAILED DESCRIPTION:
Involving caregivers in a pain coping skills protocol is likely to optimize treatment outcomes in several ways.

First, people with dementia (PWD) are likely to have difficulty learning and remembering pain coping skills; training the caregiver to coach the patient in the use of the skills is likely to improve the patients' acquisition and ongoing use of learned skills.

Second, caregiver involvement in pain coping skills training may increase their understanding of how to gauge how much pain the PWD is experiencing and the impact of pain management strategies. This understanding is increasingly important as the patient's disease progresses, and s/he is less able to report pain verbally.

Third, caregiver-assisted pain management training may enhance caregivers' self-confidence for managing the patient's pain.

Finally, by participating in the pain coping skills training protocol, caregivers may learn coping skills (such as relaxation) that can help them manage the stress associated with caring for a PWD and pain which can be significant.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Mild or moderate dementia
* Pain on most days for at least 3 months that interferes with function
* Living at home (non-institutional)
* Age ≥ 50
* English Speaking

Caregivers:

* Provides on average at least 4 hours/day of care/assistance to the patient
* Age ≥ 18
* English Speaking

Exclusion Criteria:

Patient and caregivers

* Lacking capacity for interview or unable to provide informed consent/assent.
* Visual or hearing impairments or severe behavioral problems that preclude participation.
* Too sick to participate.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-13 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Client Satisfaction Questionnaire | Post-intervention (approximately 8 weeks)
  Caregiver completes. Score range: 1-4; higher score indicates better outcome

SECONDARY OUTCOMES:
Quality of life in Alzheimer's Disease Caregiver version and Patient version | Baseline and post-intervention (approximately 8 weeks)
  Patient and Caregiver will complete Patient QOL. Score range: 13-52; higher score indicates better outcome
Brief Pain Inventory-Interference Items | Baseline and post-intervention (approximately 8 weeks)
  Patient and Caregiver will complete Patient pain interference. Score range: 0-10; higher score indicates worse outcome
Caregiver Self-Efficacy in Pain Management | Baseline and post-intervention (approximately 8 weeks)
  Caregiver will complete caregiver self-efficacy. Score range: 0-10; higher score indicates better outcome
Numeric pain scale & verbal descriptor | Baseline and post-intervention (approximately 8 weeks)
  Patient will complete patient pain intensity. Score range: 0-19; higher score indicates worse outcome
Checklist of nonverbal pain indicators | Baseline and post-intervention (approximately 8 weeks)
  Caregiver will complete patient pain intensity. Score range: 0-10; higher score indicates worse outcome
Zarit burden interview | Baseline and post-intervention (approximately 8 weeks)
  Caregivers will complete caregiver burden. Score range: 0-88; higher score indicates worse outcome
Caregiver appraisal-satisfaction scale | Baseline and post-intervention (approximately 8 weeks)
  Caregiver will complete caregiver satisfaction. Score range: 0-10; higher score indicates worse outcome
Neuropsychiatric inventory | Baseline and post-intervention (approximately 8 weeks)
  Caregiver will complete patient neuropsychiatry behaviors. Score range: 0-144; higher score indicates worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Laura Porter, Ph.D, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No